CLINICAL TRIAL: NCT04240912
Title: Confirmation of Epidural Catheter Location by Epidural Pressure Waveform Recordings by the CompuFlo® Cath-Checker System in Laboring Women.
Brief Title: Epidural Pressure Waveform Recordings by the CompuFlo® Cath-Checker System
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Other Study IDs: EESOA4
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia, Epidural
Keywords: Epidural labor analgesia; Epidural catheter assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: CompuFlo Epidural Computer Controlled System — The CompuFlo Epidural Instrument allows the objective identification of the epidural space by pressure measurement at the needle tip and consequently enables the physician to perform epidural anesthesia and epidural injections using standard methods. However, for the purpose of this study the instrument will be used only as a monitor to detect the occurrence of EPW.
  The CompuFlo Epidural Computer Controlled Anesthesia System has received a CE mark in the European Union and it received 510(k) clearance from the FDA in June 2017.

SUMMARY:
The purpose of this single arm, open label study will be to evaluate whether the dwell time of the epidural catheter, patients' position, the presence of active labor contractions and the priming volume of the epidural catheter may affect the sensitivity and specificity of CompuFlo to detect epidural pulse waveforms (EPW) to assess the correct placement of the catheter in the epidural space.

DETAILED DESCRIPTION:
The purpose of this single arm, open label study will be to evaluate whether the dwell time of the epidural catheter, patients' position, the presence of active labor contractions and the priming volume of the epidural catheter may affect the sensitivity and specificity of CompuFlo to detect epidural pulse waveforms (EPW) to assess the correct placement of the catheter in the epidural space.

The primary objective will be the correlation between the appearance of EPW recorded by the CompuFlo and the correct placement of the epidural catheter as assessed by the occurrence of adequate bilateral labor analgesia.

Secondary objectives will be the effects of the dwell time of the epidural catheter, patients' position, the presence of active labor contractions and the priming volume of the epidural catheter on the EPW.

The study will enroll consecutive parturients in active labor who have received effective epidural labor analgesia with an epidural catheter. After epidural catheter priming, the occurrence or the absence of EPW will be investigated.

Endpoints (quantitative measurements required by the objectives)

Primary end points:

1. appearance and recording of EPW by using the CompuFlo instrument.
2. absence of EPW in case of inadequate analgesia, intravascular placement or unilateral analgesia 3) successful analgesia, defined as the occurrence of a visual analogue pain score less than 10/100 during the study period

Secondary end points:

* time from the last epidural bolus and the EPW recordings
* EPW recordings between uterine contractions and at the apex of a uterine contraction
* EPW recordings when the patient is supine or in left lateral decubitus
* EPW recordings during 10 sec Valsalva maneuver
* priming volume of saline necessary to detect EPW (5,10,15,20 ml)

Tertiary end points:

* epidural actual pressure (mmHg)
* EPW disappearance or absence during catheter removal or during ineffective analgesia

ELIGIBILITY:
Inclusion Criteria:

* healthy women in active labor who received epidural analgesia

Exclusion Criteria:

* healthy women in active labor who received ineffective epidural analgesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — laboring women
Study Population: healthy women in active labor who received epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
occurrence of epidural pulse waves (EPW) | up to 5 minutes
  The occurrence of EPW recorded by the CompuFlo in working epidural catheters (epidural catheter which have produced epidural block)

SECONDARY OUTCOMES:
patient position | up to 10 minutes
  Whether patients' position (sitting or left lateral decubitus) affects the presence/absence of epidural pulse wave and/or its amplitude
uterine contractions | up to 10 minutes
  Whether the presence/absence of epidural pulse wave and/or its amplitude changes during uterine contraction in laboring women
valsalva | up to 10 minutes
  Whether the presence/absence of epidural pulse wave and/or its amplitude changes during the Valsava maneuvre in laboring women

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Città di Roma Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capogna G, Camorcia M, Coccoluto A, Micaglio M, Velardo M. Experimental validation of the CompuFlo(R) epidural controlled system to identify the epidural space and its clinical use in difficult obstetric cases. Int J Obstet Anesth. 2018 Nov;36:28-33. doi: 10.1016/j.ijoa.2018.04.008. Epub 2018 May 4. PMID 29914784
- [Background] Vaira P, Camorcia M, Palladino T, Velardo M, Capogna G. Differentiating False Loss of Resistance from True Loss of Resistance While Performing the Epidural Block with the CompuFlo(R) Epidural Instrument. Anesthesiol Res Pract. 2019 Feb 3;2019:5185901. doi: 10.1155/2019/5185901. eCollection 2019. PMID 30863447
- [Background] Gebhard RE, Moeller-Bertram T, Dobecki D, Peralta F, Pivalizza EG, Rupasinghe M, Ilic S, Hochman M. Objective Epidural Space Identification Using Continuous Real-Time Pressure Sensing Technology: A Randomized Controlled Comparison With Fluoroscopy and Traditional Loss of Resistance. Anesth Analg. 2019 Nov;129(5):1319-1327. doi: 10.1213/ANE.0000000000003873. PMID 31237571
- [Background] Al-Aamri I, Derzi SH, Moore A, Elgueta MF, Moustafa M, Schricker T, Tran DQ. Reliability of pressure waveform analysis to determine correct epidural needle placement in labouring women. Anaesthesia. 2017 Jul;72(7):840-844. doi: 10.1111/anae.13872. Epub 2017 Apr 17. PMID 28419420